CLINICAL TRIAL: NCT03944928
Title: ThOracic Ultrasound in Idiopathic Pulmonary Fibrosis Evolution
Acronym: TOUPIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19-TOUPIE
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Lung ultrasound; B lines; Pleural irregularity
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lung ultrasound — For each usual consultation every 3 months, the patient will have clinical examination and pulmonary function tests (CPI score). Thoracic ultrasound will be made during the consultation (M0, M3, M6, M9 and M12). The presence, gravity and localisation of each ultrasound sign will be described. CT-scan data will be collected in the 3 months before the start of the study and during the study. To be enrolled in the study does not change to the usual follow-up.
  For the thoracic ultrasound, a convex probe will be used (1 to 5 MHz). Patient will be layed down in a right lateral prone position then left. Thoracic ultrasound will be timed, saved and anonymized. 14 intercostal spaces will be explored by experimented operator.
  The records will be seen a second time by same operator then a second operator. this will measured interoperator and intraoperator variability.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is one of the most common chronic idiopathic fibrotic interstitial lung disease (ILD). IPF is an evolving disease that requires regular follow-up through clinical examination, respiratory functional investigations and thoracic CT. Thoracic CT is necessary for the follow-up, usually performed yearly, and in case of deterioration of respiratory function. The disadvantages to its realization are the repeated irradiation, the cost, the accessibility, and sometimes the difficulties of realization related to the supine position.

Several signs of thoracic ultrasound have been described in ILD, including the number of B lines, the irregularity of the pleural line, and the thickening of the pleural line. Cross-sectional studies have correlated the intensity of these signs with the severity of fibrosis lesions on chest CT in patients with ILD, including IPF. However, no studies have prospectively described the evolution of ultrasound signs in the same IPF patient, or their correlation to clinical, functional and CT scan evolution.

The hypothesis is that thoracic ultrasound is a relevant tool to highlight the evolution of pulmonary lesions in IPF.

The main objective is to show with thoracic ultrasound an increase in one or more of the ultrasound signs: line B score, pleural line irregularity score, and pleural line thickness during the follow-up of patient with IPF.

The study will enroll patients with a validated diagnosis of IPF in a multidisciplinary staff. At each follow-up visit, patients will have a clinical examination, pulmonary functional test and thoracic ultrasound. The CT data collected will include the last thoracic CT performed in the 3 months before the inclusion and those performed during the patient's participation. The presence, location and severity of ultrasound signs, will be recorded for each patient during successive reassessments and correlation to clinical, functional and CT scan evolution will be made.

This study will add significant knowledge in the study of ultrasound signs evolution in patients with IPF. If there is a correlation with the clinical or CT scores, it will be possible to carry over the realization of the CTs to limit the irradiation of the patients. Conversely, early detection of worsening ultrasound signs may lead to faster therapeutic adjustments to limit the extent of irreversible fibrotic lesions.

DETAILED DESCRIPTION:
- Clinical and scientic background Interstitial lung disease (ILD) is defined by an inflammatory, often fibrotic, and diffuse process, predominant in the pulmonary interstitium. Idiopathic pulmonary fibrosis (IPF) is one of the most common chronic idiopathic fibrotic interstitial lung disease. IPF is an scalable disease that requires regular follow-up through clinical examination and respiratory functional investigations. A thoracic CT scan is usually performed annually in the absence of exacerbation. CT scan is essential for initial diagnosis and follow-up, especially in case of deterioration of respiratory function. The main disadvantages to its realization are the repeated irradiation, the cost, the accessibility, and sometimes the difficulties of realization related to the supine position and the maintenance of a prolonged apnea in patients with severe dyspnea.

For several years, the semiology of interstitial lung diseases has been enriched by the description of several signs of thoracic ultrasound, including the number of B lines, the irregularity of the pleural line, and the thickening of the pleural line. Several cross-sectional studies have correlated the intensity of these signs with the severity of fibrosis lesions on chest CT in patients with ILD, including IPF. However, no studies have prospectively described the evolution of ultrasound signs in the same IPF patient, or their correlation to clinical, functional and CT evolution.

The hypothesis is that thoracic ultrasound is a relevant tool to highlight the evolution of pulmonary lesions in IPF.

* Objective of the study: The main objective is to show with thoracic ultrasound an increase in one or more of the ultrasound signs: line B score, pleural line irregularity score, and pleural line thickness during the follow-up of patient with IPF. The secondary objectives are to evaluate the reproducibility of the measurements of the pulmonary ultrasound signs, to evaluate the association between the severity of each pulmonary ultrasound sign and the severity of the clinical, functional and CT scores and to evaluate the association between the measurement of each ultrasound sign made during a standard protocol exploring 14 intercostal spaces and a simplified protocol exploring 6 intercostal spaces.
* Design: This is a prospective, multicenter, non-interventional, prospective study evaluating patients followed for IPF at the University Hospital of Tours and the Hospital of Orléans, France.

Number of participants: 30

- Interventions and analysis: The study will enroll patients with a validated diagnosis of IPF in a multidisciplinary staff. For each patient included, study duration will be 12 months. At each follow-up visit, patients will have a clinical examination, pulmonary functional test and thoracic ultrasound. The CT data collected will include the last thoracic CT performed in the 3 months before the inclusion and those performed during the patient's participation.

Thoracic ultrasonography will be performed on D0, M3, M6, M9 and M12. It will occur during the follow-up consultation carried out as part of usual care. Thus, inclusion in the study does not change the usual rhythm of consultations or complementary examinations (pulmonary functional tests and thoracic CT scan) in the care of the patient.

A convex probe (1 to 5 MHz) will be used. The patient will be placed in right lateral decubitus then left. Thoracic ultrasonography will be timed, recorded and anonymized. It will be practiced by experienced operators and according to a validated protocol allowing the exploration of 14 intercostal spaces. The recording loops will be read over later by the operator himself and then by a second operator to evaluate the intra- and inter-operator variability respectively.

The presence, location and severity of ultrasound signs, will be recorded for each patient during successive reassessments and correlation to clinical, functional and CT scan evolution will be made.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years-old
* diagnosis of IPF validated in a multidisciplinary consultation meeting (RCP) according to French recommendations

Exclusion Criteria:

* pregnant or lactating women
* exacerbation of fibrosis on inclusion
* right or left heart aggravation on inclusion
* evolutive pulmonary infectious disease
* other forms of diffuse interstitial lung disease
* opposition to the data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with idiopathic pulmonary fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Change of the B-line score from inclusion to 12 months | Inclusion, 12 months
  number of line
Change of pleural line irregularity from inclusion to 12 months | Inclusion, 12 months
  Percentage
Change of pleural line thickness from inclusion to 12 months | Inclusion, 12 months
  in millimeters

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHR Orleans, Orléans
  - Pulmonology Department, University Hospital, Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Legue S, Marchand-Adam S, Plantier L, Bayeh BA, Morel H, Mangiapan G, Flament T. ThOracic Ultrasound in Idiopathic Pulmonary Fibrosis Evolution (TOUPIE): research protocol of a multicentric prospective study. BMJ Open. 2021 Mar 25;11(3):e039078. doi: 10.1136/bmjopen-2020-039078. PMID 33766834